CLINICAL TRIAL: NCT02961062
Title: A Randomized, Vehicle-controlled, Subject and Investigator-masked, Proof-of-concept Study to Evaluate the Use of Topical Ocular SAF312 in the Treatment of Postoperative Ocular Pain in Patients Undergoing Photorefractive Keratectomy (PRK) Surgery
Brief Title: Study of SAF312 as an Eye Drop for Treatment of Eye Pain Following Photorefractive Keratectomy (PRK) Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSAF312X2201
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Results first posted 2019-04-11 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Ocular Pain After PRK Surgery
Keywords: ocular pain; photorefractive keratectomy (PRK); SAF312; corneal epithelial defect
MeSH Terms: conditions — Eye Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence 1 (Experimental)
  Interventions: Drug: SAF312; Drug: Placebo
- Treatment Sequence 2 (Placebo Comparator)
  Interventions: Drug: SAF312; Drug: Placebo

INTERVENTIONS:
Drug: SAF312
Drug: Placebo

SUMMARY:
The purpose of this study is to determine if SAF312 eye drops have an adequate safety and efficacy profile to justify further clinical development for the treatment of ocular pain associated with corneal epithelial defect such as after photorefractive keratectomy (PRK) surgery

ELIGIBILITY:
Inclusion Criteria:

* Normal eye exam except for refractive error at baseline.
* Myopia should not exceed -4.00 Diopters (sphere) and 3.00 diopters of astigmatism, with spherical equivalent not higher than -4.50, confirmed by manifest refraction at baseline.

Exclusion Criteria:

* Monocular patient (including amblyopia) or best corrected visual acuity score worse than 20/80 (Snellen) or 55 letters (EDTRS), at baseline.
* Any systemic or ocular disease that might affect wound healing (such as severe rheumatoid arthritis or diabetes or history of keloid formation) or a history of ocular trauma, uveitis, infection, or inflammation in the 6 months prior to baseline.
* Previous refractive or corneal surgery (such as LASIK, PRK, radial keratotomy, pterygium removal, corneal transplantation).
* Chronic pain of any etiology or any significant illness which has not resolved within two (2) weeks prior to initial dosing.

Other inclusion and exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - Novartis Investigative Site, Chevy Chase, Maryland
  - Novartis Investigative Site, Sioux Falls, South Dakota
  - Novartis Investigative Site, Draper, Utah
  - Novartis Investigative Site, Norfolk, Virginia

REFERENCES:
- [Derived] Mangwani-Mordani S, Goodman CF, Galor A. Novel Treatments for Chronic Ocular Surface Pain. Cornea. 2023 Mar 1;42(3):261-271. doi: 10.1097/ICO.0000000000003193. Epub 2022 Dec 19. PMID 36729473
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=436

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 40 patients were randomized in a 1:1 ratio to two treatment sequences: SAF312 followed by Vehicle, or Vehicle followed by SAF312.
Pre-assignment Details: Bilateral crossover design: A crossover design was utilized in order to decrease the inter-patient variability due to different pain tolerance in different individuals.
Groups:
- Treatment Sequence 1: Vehicle/SAF312
- Treatment Sequence 2: SAF312 / Vehicle
Period: Overall Study
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (10.77) | 33.7 (8.94) | 34.0 (9.78)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  male | 11 | 10 | 21
  female | 9 | 10 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    white | 18 | 17 | 35
    asian | 2 | 1 | 3
    Black | 0 | 1 | 1
    multiple | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    non hispanic latino | 19 | 18 | 37
    hispanic latino | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Pre-dose Pain Assessment
Description: VAS pain severity scale pre-dose, 6 hours post-operatively. The Visual Analog Scale (VAS) is a commonly used measurement of pain, discomfort, that goes from 0 meaning no pain to 100 meaning worst imaginable pain
Time Frame: 6 hours
Population: Primary PD Analysis set
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- SAF312: treatment participants from both sequences
- Vehicle: comparator participants from both sequences
Arm/Group | SAF312 | Vehicle
Number analyzed (Participants) | 40 | 40
score on a scale | 34.63 (4.05) | 45.76 (4.10)
Statistical Analysis 1: Comparison: SAF312 vs Vehicle; Test type: Superiority; p = 0.005, Kenward-Roger method; Mean Difference (Final Values) = -11.1, 90% CI 2-sided [-17.54 to -4.71], Standard Error of Mean 0

2. Primary Outcome: Average Ocular Pain VAS Assessments
Description: VAS pain severity scale from the first post-operative assessment to pre-dose 12 hours post-operative assesment The Visual Analog Scale (VAS) is a commonly used measurement of pain, discomfort, that goes from 0 meaning no pain to 100 meaning worst imaginable pain
Time Frame: 12 hours
Population: Primary PD Analysis set
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SAF312 | Vehicle
Number analyzed (Participants) | 40 | 40
score on a scale | 30.90 (4.07) | 39.47 (4.11)
Statistical Analysis 1: Comparison: SAF312 vs Vehicle; Test type: Superiority; p = 0.017, Kenward-Roger method; Median Difference (Final Values) = -8.56, 90% CI 2-sided [-14.29 to -2.83], Standard Error of Mean 3.37

3. Secondary Outcome: Incidence of and Amount of Rescue Oral Analgesics (Number of Participants Who Did Not Use Oral Rescue Medication)
Description: Summary of oral rescue medication use incidence (number of patients who DID NOT use oral rescue medication)
Time Frame: 6,12, 24, 48 and 72 hours post-operatievly
Population: Secondary PD analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | SAF312 | Vehicle
Number analyzed (Participants) | 40 | 40
Participants
  0-6 hours post-operatively | 23 | 19
  0-12 hours post-operatively | 19 | 16
  0-24 hours post-operatively | 16 | 12
  0-48 hours post-operatively | 11 | 11
  0-72 hours post-operatively | 11 | 11

4. Secondary Outcome: VAS Pain Assessments
Description: VAS pain assessment during the first 72 hours post-operatively. VAS pain severity scale from the first post-operative assessment to pre-dose 12 hours post-operative assesment The Visual Analog Scale (VAS) is a commonly used measurement of pain, discomfort, that goes from 0 meaning no pain to 100 meaning worst imaginable pain
Time Frame: 72 hours
Population: Primary PD Analysis set
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SAF312 | Vehicle
Number analyzed (Participants) | 40 | 40
score on a scale | 5.13 (4.05) | 3.58 (4.10)

5. Secondary Outcome: Plasma Concentration of SAF312
Description: C Max
Time Frame: day1, day 4
Population: PK Analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SAF312 | Vehicle
Number analyzed (Participants) | 40 | 40
ng/mL
  day 1: number analyzed (Participants) | 34 | 0
  day 1 | 0.454 (0.227) |
  day 4: number analyzed (Participants) | 33 | 0
  day 4 | 2.40 (1.53) |

ADVERSE EVENTS:
Time Frame: approximately 15 months
Groups:
- Vehicle: Vehicle
Arm/Group | SAF312 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 8/40 | 5/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAF312 (N=40) | Vehicle (N=40)
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Corneal infiltrates (Eye disorders) | 0 | 1
Corneal opacity (Eye disorders) | 1 | 1
Punctate keratitis (Eye disorders) | 1 | 1
Vitreous detachment (Eye disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT02961062/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT02961062/SAP_001.pdf